CLINICAL TRIAL: NCT05853328
Title: Benign Peripheral Paroxysmal Positional Vertigo (BPPV): Comparison of the Epley Maneuver With the So-called SémontPLUS Liberation Maneuver
Brief Title: Comparison of EM and SM+ Maneuvers in Patients With BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Michael Strupp, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-072
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: BPPV
Keywords: Benign paroxysmal positional vertigo; SemontPLUS maneuver; Epley maneuver
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of two test groups. After being randomized to the SM+ arm or the EM arm, patients will receive one initial maneuver from a physician, then subsequently performe self-maneuvers at home three times in the morning, three times at noon and three times in the evening.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epley Maneuver (Active Comparator): The SOC therapy for this patient population is Physical Therapy. No medication or medical device therapy was included. In addition to SOC, patients in this arm were allocated to Epley Maneuver. The first treatment maneuver was performed once by a physician according to the assigned treatment group. The patient simultaneously received verbal instructions on how to perform the maneuver. Fifteen minutes after the first diagnostic maneuver, a second diagnostic maneuver was carried out in order to evaluate the effect of a single maneuver.
  For the self-maneuvers, patients received written instructions with figures on how to perform the EM independently in a home environment. For the self-maneuver at home, the modified Epley self-maneuver was done by the patient with a pillow under the shoulders.
  The frequency at home was three times in the morning, three times at noon, and three times in the evening, i.e., nine times per day.
  Interventions: Procedure: Epley Maneuver
- SemontPLUS Maneuver (Active Comparator): The SOC therapy for this patient population is Physical Therapy. No medication or medical device therapy was included. In addition to SOC, patients in this arm were allocated to the SemontPLUS Maneuver. The first treatment maneuver was performed once by a physician according to the assigned treatment group. For the SM+, the angle of the 60° overextended head and body was measured by an inclinometer application. The patient simultaneously received verbal instructions on how to perform the maneuver. Fifteen minutes after the first diagnostic maneuver, a second diagnostic maneuver was carried out in order to evaluate the effect of a single maneuver.
  For the self-maneuvers, patients received written instructions with figures on how to perform the SM+ independently in a home environment.
  The frequency at home was three times in the morning, three times at noon, and three times in the evening, i.e., nine times per day.
  Interventions: Procedure: SemontPLUS maneuver

INTERVENTIONS:
Procedure: Epley Maneuver — The patient is sitting with both feet on the table or bed with the head looking forward. Subsequently, they let themselves fall backwards with a pillow under the shoulder and the head is turned 45° to the right. They stay in this position for 30 seconds. Afterwards, they turn the head quickly 90° to the left side followed by a turn of the whole body to the left so that their nose is pointing at the floor. They stay in this position for another 30 seconds.
  Subsequently, the patients sit themselves up with the head still turned 45° to the left. They can help themselves by using both arms. After a few seconds, they can turn the head slowly back to the neutral position facing forward.
  Arms: Epley Maneuver
Procedure: SemontPLUS maneuver — The patients first turn head 45° to the left. Then they extend the right arm and subsequently move the whole body by 150°+ to the right side. This position is kept for 60 seconds. Subsequently, patients move their whole body by 240° towards the non-affected side. Finally, after another 60 seconds, the patient sits up for another 60 sec.
  Arms: SemontPLUS Maneuver

SUMMARY:
Objective of this prospective randomized treatment trial is to compare the effectiveness of the SemontPLUS (SM+) with the Epley maneuver (EM) for the therapy of posterior canal benign paroxysmal positional vertigo canalolithiasis (pcBPPV).

DETAILED DESCRIPTION:
BPPV is the second most common form of vertigo. Reported prevalence ranges from 10 to 140 per 100,000 and lifetime prevalence is at least 2.4%; prevalence of 9-11% have been found in a population older than 75 years.

The leading symptom is recurrent attacks of spinning vertigo, each triggered by changes in position relative to gravity and lasting from seconds to one minute. The cause is usually freely moving otoconia in the posterior arcuate canal (so-called canalolithiasis); the horizontal canal is affected much less frequently. In 70% of patients there is a spontaneous remission within days. In case of persistence, about 95% of patients can be successfully treated with so-called freeing maneuvers, e.g., the Sémont maneuver. However, this often requires 20 to 30 maneuvers over several days.

Based on

1. our own biophysical studies, which we performed together with colleagues from Switzerland on a mechanical model of positional vertigo and which show that theoretically 24 the effectiveness of the Sémont maneuvers can be increased by changing the positional angle by 30° in the so-called step two of the positional maneuvers, as well as
2. an analysis of the comparison of the conventional Sémont maneuver with the so-called SémontPLUS maneuver, which shows that the mean time to freedom from symptoms for the Sémont maneuver is 3.9 days and only 2.3 days for the SémontPLUS maneuver (p<0.05), the efficacy of the Epley maneuver will be compared with the SemontPLUS maneuver in a parallel group design.

The primary endpoint is the duration, i.e., days ("mornings") until freedom from symptoms with continuation of the two maneuvers in the following days, three times in the morning, at noon and in the evening. This is assessed by the patient's statements that he/she can still induce rotational vertigo or not during the positioning maneuvers to the affected side performed by him/herself.

ELIGIBILITY:
Inclusion Criteria:

* Subject (≥ 18 years of age) meets diagnostic criteria for the current presence of BPPV of a posterior arcuate duct (8):

History: rotary vertigo attacks triggered by head or body position change. Duration: < 1 minute, associated with nausea, vomiting, oscillopsia

Findings: When positioned to the affected ear: torsional and vertically to the forehead beating, exhaustive nystagmus with crescendo-decrescendo-like course.

Exclusion Criteria:

* Subjects not capable of giving consent
* Respondent does not want therapy for BPPV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Number of days until no positional vertigo could be induced | 28 days
  Patients had to document whether they could provoke positional vertigo every morning. The primary endpoint was the number of days until no positional vertigo could be induced on three subsequent mornings.

SECONDARY OUTCOMES:
Effect of the single maneuver performed by the physician. | 28 days
  How many patients in both treatment groups become vertigo and nystagmus-free after a single performance of the allocated treatment maneuver performed by a physician.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Strupp, Principal Investigator — LMU University
Locations (3):
- Department of ENT, AZ Sint-Jan Brugge-Oostende AV, Ostend, Flanders, Belgium
- Department of Neurology, Ludwig Maximilian University, Munich, Bavaria, Germany
- Department of ENT, University of Siena, Siena, Italy

REFERENCES:
- [Derived] Strupp M, Mandala M, Vinck AS, Van Breda L, Salerni L, Gerb J, Bayer O, Mavrodiev V, Goldschagg N. The Semont-Plus Maneuver or the Epley Maneuver in Posterior Canal Benign Paroxysmal Positional Vertigo: A Randomized Clinical Study. JAMA Neurol. 2023 Aug 1;80(8):798-804. doi: 10.1001/jamaneurol.2023.1408. PMID 37358870